CLINICAL TRIAL: NCT06480981
Title: A Randomized, Double-blind, Placebo-controlled Trial to Evaluate Multiple Dose Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Ascending Doses of Noribogaine in Healthy Volunteers.
Brief Title: Multiple Ascending Dose Noribogaine PK/PD in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DemeRx NB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: DMX-NB-001
Record Dates: First submitted 2024-06-19; First posted 2024-07-01 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — noribogaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Noribogaine 20mg (Experimental): 1 x Noribogaine 10mg capsule twice daily
  Interventions: Drug: Noribogaine
- Noribogaine 40mg (Experimental): 1 x Noribogaine 20mg capsule twice daily
  Interventions: Drug: Noribogaine
- Noribogaine 60mg (Experimental): 1 x Noribogaine 10mg capsule and 1 x Noribogaine 20mg capsule twice daily
  Interventions: Drug: Noribogaine
- Noribogaine 80mg (Experimental): 2 x Noribogaine 20mg capsule twice daily
  Interventions: Drug: Noribogaine

INTERVENTIONS:
Drug: Noribogaine — Noribogaine capsules

SUMMARY:
This trial will be a randomised, double-blind, sequential-group, multiple-dose, placebo-controlled, dose escalation trial to characterise the pharmacokinetics (PK), pharmacodynamics (PD) and safety of noribogaine in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written, personally signed, and dated informed consent.
* Healthy male and female participants between the ages of 18 to 45 inclusive.
* BMI 18 - 30 kg/m2.
* Non- or ex-smoker.
* Normal ECG findings i.e. QTcF interval ≤ 450 ms and normal morphology that would permit accurate assessment of the QT interval.
* Participants must agree to use highly

Exclusion Criteria:

* History of, or concurrent clinically significant cardiovascular, dysautonomia, gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic or psychiatric, or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the participant or impact the validity of the study.
* Family history in first degree relatives for unknown and/or known arrhythmia-related cardiac events, cardiomyopathy, syncope, long QT syndrome, Brugada's syndrome, sudden death attributed to cardiac causes, and familial cardiac channelopathies.
* Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with interpretation of QTc interval changes.
* Previous or current alcohol, or other drug dependence.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2025-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorg Taubel, Principal Investigator — Richmond Pharmacology
Locations (1):
- Richmond Pharmacology, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited at a single dedicated site - Richmond Pharmacology.
Pre-assignment Details: All participants enrolled in the study were assigned to a treatment group.
Groups:
- Placebo: Placebo capsules twice daily
Period: Overall Study
Arm/Group | Noribogaine 20mg | Noribogaine 40mg | Noribogaine 60mg | Noribogaine 80mg | Placebo
Started | 10 | 12 | 12 | 9 | 12
Completed | 10 | 12 | 12 | 9 | 12
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Noribogaine 20mg | Noribogaine 40mg | Noribogaine 60mg | Noribogaine 80mg | Placebo | Total
Number analyzed (Participants) | 10 | 12 | 12 | 9 | 12 | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.0 (5.14) | 28.7 (7.6) | 31.1 (6.96) | 29.1 (4.91) | 29.3 (5.5) | 29.1 (6.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 9 | 3 | 4 | 20
  Male | 9 | 9 | 3 | 6 | 8 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 4 | 0 | 1 | 4 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 6 | 7 | 4 | 21
  White | 2 | 5 | 5 | 1 | 3 | 16
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 1 | 0 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 10 | 12 | 12 | 9 | 12 | 55
BMI [Mean (Standard Deviation); unit: kg/m2] | 22.5 (3.1) | 23.9 (2.36) | 23.2 (2.45) | 24.6 (3.01) | 24.9 (2.35) | 23.8 (2.68)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics Cmax Day 1
Description: Determination of maximum plasma concentration of noribogaine
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Noribogaine 20mg | Noribogaine 40mg | Noribogaine 60mg | Noribogaine 80mg
Number analyzed (Participants) | 10 | 12 | 12 | 9
ng/ml | 10.4 (3.26) | 22.7 (8.47) | 39.5 (8.27) | 45.2 (10.5)

2. Primary Outcome: Pharmacokinetics Cmax Day 8
Description: Determination of maximum plasma concentration of noribogaine
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Noribogaine 20mg | Noribogaine 40mg | Noribogaine 60mg | Noribogaine 80mg
Number analyzed (Participants) | 10 | 12 | 12 | 9
ng/ml | 28.7 (13.1) | 45.5 (19.7) | 91.9 (30.6) | 113 (27.9)

3. Primary Outcome: Pharmacokinetics Tmax Day 1
Description: Determination of the time to reach the maximum plasma concentration of noribogaine
Time Frame: Day 1
Measure: Median (Full Range); unit: hours
Arm/Group | Noribogaine 20mg | Noribogaine 40mg | Noribogaine 60mg | Noribogaine 80mg
Number analyzed (Participants) | 10 | 12 | 12 | 9
hours | 4.01 [2.5 to 8] | 2.75 [1.5 to 8.03] | 3.27 [2 to 8.07] | 3.50 [1.5 to 8.07]

4. Primary Outcome: Pharmacokinetics Tmax Day 8
Description: Determination of the time to reach the maximum plasma concentration of noribogaine
Time Frame: Day 8
Measure: Median (Full Range); unit: hours
Arm/Group | Noribogaine 20mg | Noribogaine 40mg | Noribogaine 60mg | Noribogaine 80mg
Number analyzed (Participants) | 10 | 12 | 12 | 9
hours | 3.5 [1.5 to 4.0] | 1.87 [1.0 to 3.53] | 2.53 [1.5 to 4.0] | 3.0 [1.0 to 4.0]

5. Primary Outcome: Pharmacokinetics AUC0-t Day 1
Description: Determination of the area under the plasma concentration-time curve from time 0 to t of noribogaine
Time Frame: Day 1
Population: Insufficient datapoints to determine AUC for the missing participants.
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | Noribogaine 20mg | Noribogaine 40mg | Noribogaine 60mg | Noribogaine 80mg
Number analyzed (Participants) | 6 | 8 | 9 | 5
ng·h/mL | 87.8 (40.1) | 196 (48.0) | 335 (92.2) | 414 (72.6)

6. Primary Outcome: Pharmacokinetics AUC0-t Day 8
Description: Determination of the area under the plasma concentration-time curve from time 0 to t of noribogaine
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: ng h/ml
Arm/Group | Noribogaine 20mg | Noribogaine 40mg | Noribogaine 60mg | Noribogaine 80mg
Number analyzed (Participants) | 10 | 12 | 12 | 9
ng h/ml | 289 (152) | 429 (215) | 847 (329) | 1030 (275)

7. Primary Outcome: Pharmacokinetics AUC0-infinity Day 8
Description: Determination of the area under the plasma concentration-time curve from time 0 to infinity of noribogaine
Time Frame: Day 8
Population: Insufficient datapoints to determine AUC for missing participant.
Measure: Mean (Standard Deviation); unit: ng h/ml
Arm/Group | Noribogaine 20mg | Noribogaine 40mg | Noribogaine 60mg | Noribogaine 80mg
Number analyzed (Participants) | 9 | 12 | 12 | 9
ng h/ml | 934 (675) | 974 (679) | 2200 (1330) | 2550 (1210)

8. Primary Outcome: Pharmacokinetics t1/2 Day 1
Description: Determination of elimination half-life (t1/2) of noribogaine
Time Frame: Day 1
Population: Insufficient datapoints to calculate Thalf.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Noribogaine 20mg | Noribogaine 40mg | Noribogaine 60mg | Noribogaine 80mg
Number analyzed (Participants) | 6 | 6 | 9 | 4
hours | 13.8 (4.2) | 10.5 (4.52) | 9.59 (2.38) | 11.5 (3.16)

9. Primary Outcome: Pharmacokinetics t1/2 Day 8
Description: Determination of elimination half-life (t1/2) of noribogaine
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Noribogaine 20mg | Noribogaine 40mg | Noribogaine 60mg | Noribogaine 80mg
Number analyzed (Participants) | 10 | 12 | 12 | 9
hours | 23.0 (11.3) | 14.0 (4.34) | 28.4 (19.7) | 25.4 (12.1)

ADVERSE EVENTS:
Time Frame: From baseline until end of follow-up, up to 15 days.
Arm/Group | Noribogaine 20mg | Noribogaine 40mg | Noribogaine 60mg | Noribogaine 80mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12 | 0/12 | 0/9 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/12 | 0/9 | 0/12
Other Adverse Events (participants affected / at risk) | 4/10 | 8/12 | 11/12 | 9/9 | 8/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Noribogaine 20mg (N=10) | Noribogaine 40mg (N=12) | Noribogaine 60mg (N=12) | Noribogaine 80mg (N=9) | Placebo (N=12)
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Vascular access site bruising (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 2 | 6 | 7 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 6 | 9 | 5 | 8
Dizziness postural (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Presyncope (Vascular disorders) | 1 | 2 | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT06480981/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-19): https://cdn.clinicaltrials.gov/large-docs/81/NCT06480981/SAP_001.pdf